CLINICAL TRIAL: NCT02912234
Title: Effect of Clarithromycin on the Pharmacokinetics of Apixaban in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CV185-547
Record Dates: First submitted 2016-09-19; First posted 2016-09-23 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — apixaban; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apixaban and Clarithromycin (Experimental)
  Interventions: Drug: Apixaban; Drug: Clarithromycin

INTERVENTIONS:
Drug: Apixaban — Multiple-dose clarithromycin and single-dose Apixaban
Drug: Clarithromycin — Multiple-dose clarithromycin and single-dose Apixaban

SUMMARY:
This study is to evaluate the effects of multiple-dose clarithromycin on the single-dose pharmacokinetics (PK) of apixaban with parameters like Cmax, AUC(INF), and AUC(0-T).

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Target population: Healthy subjects as determined by medical history, surgical history, physical examination, vital signs, electrocardiogram (ECG), and clinical laboratory tests including coagulation parameters.
3. Subjects with body mass index of 18 to 30 kg/m2, inclusive
4. Women must not be breast feeding, have a negative serum or urine pregnancy test and must agree to follow instructions for method(s) of contraception for the duration of treatment with study treatments apixaban and clarithromycin plus 5 half-lives of study treatments apixaban and clarithromycin plus 30 days (duration of ovulatory cycle) for a total of 33 days post-treatment completion.
5. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study treatments apixaban and clarithromycin plus 5 half-lives of the study treatment plus 30 days for a total of 33 days post-treatment completion. In addition, male participants must be willing to refrain from sperm donation during this time.

Exclusion Criteria:

1. History of any significant medical illness, drug allergy including allergy to apixaban, FXa inhibitors (and/or their excipients), clarithromycin, macrolides, and/or related compounds. History of substance abuse and use of nicotine containing products and/or alcohol abuse.
2. History of coagulopathy, prolonged or unexplained clinically significant bleeding, or frequent unexplained bruising or thrombus formation, including hypermenorrhea, intra-cranial hemorrhage, family history of bleeding disorders in first degree relatives, and/or any adverse reaction to anticoagulants or antiplatelet agents that resulted in excessive bleeding.
3. History of recurrent neurological or gastrointestinal disorders, including insomnia, chronic headaches, dizziness, gastroesophageal reflux disease, cholecystectomy, gastric ulcers and/or Gilbert's syndrome.
4. History of antibiotic induced secondary infections, including candidiasis.
5. Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG, or clinical laboratory tests beyond what is consistent with the target population.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Days 1-11
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | Days 1-11
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUC(0-T)) | Days 1-11

SECONDARY OUTCOMES:
Safety endpoints include the incidence of adverse events (AEs), serious adverse events (SAEs), AEs leading to discontinuation, and death | Screening- until 30 days after discontinuation of dosing or subject's participation in the study if the last

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Ppd Development, Llc, Austin, Texas, United States

REFERENCES:
- [Derived] Garonzik S, Byon W, Myers E, Li X, Marchisin D, Murthy B. The Effects of Clarithromycin on the Pharmacokinetics of Apixaban in Healthy Volunteers: A Single-Sequence Crossover Study. Am J Cardiovasc Drugs. 2019 Dec;19(6):561-567. doi: 10.1007/s40256-019-00348-2. PMID 31030414
- See also: BMS Clinical Trial Education Resource — http://www.bms.com/studyconnect/pages/home.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx